CLINICAL TRIAL: NCT04747652
Title: Clinical Research on Advanced Warning Factors Of Respiratory Injury in Dermatomyositis
Acronym: CRAWFORD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Wenfeng Tan, Chief Physician, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: MSG-jiangsu
Record Dates: First submitted 2021-02-07; First posted 2021-02-10 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Dermatomyositis; Respiratory Injury
Keywords: Dermatomyositis; Respiratory Injury; Advanced Warning
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cell, serum or plasma, muscle and lung biopsy specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dermatomyositis (DM) is a highly heterogeneous autoimmune disease characterized by rash and myasthenia. Beside these, respiratory involvement is one of the common complications of DM. Interstitial lung disease (ILD) occur in approximately 90% of patients with DM, part of them may manifest rapidly progressive-interstitial lung disease (rp-ILD), which progresses into respiratory failure that is difficult to correct and leads to death. Early identification of rp-ILD high risk group is of great significance to improve the prognosis of patients and to conduct following clinical studies. A simple, easy, convenient and reliable diagnostic tool has not yet acquired till now.

DETAILED DESCRIPTION:
Dermatomyositis (DM) is a highly heterogeneous autoimmune disease characterized by rash and myasthenia. Beside these, respiratory involvement is one of the common complications of DM. Interstitial lung disease (ILD) occur in approximately 90% of patients with DM, part of them may manifest rapidly progressive-interstitial lung disease (rp-ILD), which progresses into respiratory failure that is difficult to correct and leads to death. Early identification of rp-ILD high risk group is of great significance to improve the prognosis of patients and to conduct following clinical studies. A simple, easy, convenient and reliable diagnostic tool has not yet acquired till now.

MSG-Jiangsu, short for Myositis Study Group-Jiangsu, was founded by department of rheumatology and immunology of eighteen tertiary hospitals. Clinical Research on Advanced Warning Factors Of Respiratory Injury in Dermatomyositis (CRAWFORD) as a multicenter observational cohort study was started at Jun 1, 2020. Our cohort plan to recruit 1,000 adult inpatients. What's more, prognostic data from these DM patients were obtained by following up for 1 year. At the same time, clinical data and auxiliary examination results of the baseline DM patients were analyzed to look for factors that are associated with outcomes. Then, regression analysis of influencing factors will help us to set up a multi-factor weighted score to forecast the prognosis of DM patients. Finally, Biological specimen from patients at baseline are used to look for biomarkers that predict prognosis by RNA-sequencing, whole exon sequencing, proteomic screening and so on.

ELIGIBILITY:
Inclusion Criteria:

* adult patients meet the diagnostic criteria for dermatomyositis of Bohan and Peter

Exclusion Criteria:

* complicated with other connective tissue diseases
* complicated with cardiovascular and respiratory disease caused by other reasons
* interstitial lung disease caused by environment and drugs
* patients with key research missing data or without informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruit inpatients from department of rheumatology and immunology of eighteen tertiary hospitals in Jiangsu province
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
death | within 12 months after disease oneset
  death caused by dermatomyositis and its related complications

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wang L, Lv C, You H, Xu L, Yuan F, Li J, Wu M, Zhou S, Da Z, Qian J, Wei H, Yan W, Zhou L, Wang Y, Yin S, Zhou D, Wu J, Lu Y, Su D, Liu Z, Liu L, Ma L, Xu X, Zang Y, Liu H, Ren T, Liu J, Wang F, Zhang M, Tan W. Rapidly progressive interstitial lung disease risk prediction in anti-MDA5 positive dermatomyositis: the CROSS model. Front Immunol. 2024 Feb 1;15:1286973. doi: 10.3389/fimmu.2024.1286973. eCollection 2024. PMID 38361940